CLINICAL TRIAL: NCT05314686
Title: Technical Validity and Clinical Feasibility of Using a Telerehabilitation System Using Advanced Telehealth Technologies
Brief Title: Telerehabilitation - Technical Validity and Clinical Feasibility
Status: Completed | Type: Observational
Sponsor: ADIR Association (Other)
Collaborators: Union des Kinésithérapeutes Respiratoires (Unknown); CogSci (Unknown); KerNel Biomedical (Industry); Groupe Havrais d'Aide aux Handicapés Respiratoires (Unknown)
Responsible Party: Sponsor
Other Study IDs: TelerehApp-Valid/Feasib
Record Dates: First submitted 2022-03-25; First posted 2022-04-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Pulmonary rehabilitation; Telerehabilitation; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Technical validity of data transmitted remotely.: The first twenty participants will participate in the step of the study aimed at assessing the technical validity of data transmitted remotely from devices connected to the telerehabilitation system.
  Interventions: Other: Five exercise sessions of forty-five minutes within the pulmonary rehabilitation centre and ten days of using a physical activity tracker.
- Clinical feasibility.: The last twenty participants will perform their pulmonary rehabilitation program at home using the telerehabilitation system over an eight-week period.
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Five exercise sessions of forty-five minutes within the pulmonary rehabilitation centre and ten days of using a physical activity tracker. — 1. Five exercise sessions of forty-five minutes within the centre on a cycle ergometer using a pulse oximetry device connected to the telerehabilitation system through Bluetooth. Data recorded in the internal memory of the pulse oximeter will be compared with those transmitted through the telerehabilitation system.
  2. Ten days of use of a physical activity tracker connected to the telerehabilitation system. Self-reported daily step count by the participants (using a standardized data sheet) will be compared with the daily step count transmitted through the telerehabilitation system.
  Groups: Technical validity of data transmitted remotely.
Other: Telerehabilitation — An eight-week program including:
  * Endurance training on a cycle ergometer (performed independently with remote monitoring or through video conference, according to the participant's preference), three times per week. Training prescription is progressively adjusted using an automated algorithm (aimed to first increase the training duration and then workload intensity).
  * Peripheral muscle strengthening using the app (the patient will be requested to reproduce different exercises after watching a video) or through video conference, three times per week (thirty minutes).
  * Daily walking with automated coaching.
  * Self management education (one to nine sessions according to each individual needs, scheduled through videoconference).
  * A self evaluation of symptoms through daily or weekly questionnaires. Different types of alert will be triggered at the center according to remote monitoring: "non-adherence", "clinical issue" during endurance exercise sessions and change in "symptoms".
  Groups: Clinical feasibility.

SUMMARY:
This prospective study will be held in two steps.

The aim of the first step is to assess the technical validity of transmitting data remotely from different devices connected to a telerehabilitation system. These will include real-time oximetry data during exercise on a cycle ergometer (heart rate and transcutaneous oxygen saturation) as well as daily step count from a commercially available physical activity tracker.

The aim of the second step of the study is to assess the clinical feasibility of using the telerehabilitation system in real life conditions (in the home environment). Briefly, participants will benefit from a eight weeks pulmonary rehabilitation program performed at home, using the telerehabilitation system. Further details about the content of the program and the outcomes are provided below.

DETAILED DESCRIPTION:
Before taking part in the study, participants will undergo an incremental cardiopulmonary exercise testing as their baseline assessment before referral to a pulmonary rehabilitation program.

Participants referred for pulmonary rehabilitation to the ADIR Association will be screened for eligibility. They will be contacted to initiate their program. During the first session, they will be offered to participate in the study.

This protocol will be held in two steps : the first step will aim to assess the clinical validity of the data transmitted remotely through the system (from two different devices) and the second step will aim to assess the clinical feasibility of using the system in the home environment.

Participant recruitment for each of these steps will be performed chronologically (the first twenty eligible participants will participate in the technical validity step of the study and the last twenty eligible participants will participate in the clinical feasibility step).

Step one: Clinical validity. The first step of the study aims to assess the clinical validity of data transmitted remotely from two devices connected to the telerehabilitation system (a. oximetry data during exercise and b. daily step count from a commercially available physical activity tracker).

1. Oxymetry data during exercise on a cycle ergometer.

   Participants who agree to participate will be trained to use the system within the pulmonary rehabilitation centre. Training includes different steps such as to turn on the tablet, to connect to the application, to start the session using the app, to synchronise the oximeter with the app, to perform the session and to validate the end of the session.

   Participants will be asked to perform five endurance exercise sessions of forty-five minutes each, over five different days, within the centre. During these sessions a connected pulsed oximeter device will record heart rate and transcutaneous oxygen saturation at a frequency of one hertz. These data will be recorded in the internal memory of the oximeter itself as well as transmitted in real-time through Bluetooth to the app. The app will transmit the data to a secured remote server through the Global System for Mobile communication network. These two datasets (those locally stored and those remotely transmitted) will be analysed and compared (proportion of artefact, data deletion, data transformation, comparability etc - see outcomes for further details).
2. Data from a physical activity tracker.

Concurrently, the same participants will be asked to wear a physical activity tracker over a ten-day period. The data (daily step count) will be automatically and daily transmitted to the app through Bluetooth and then from the app to the remote secured server. Participants will be asked to remove the sensor when going to bed and to note the number of steps displayed on the screen on a standardized data sheet.

Step two: Clinical feasibility. The aim of the second step of the study is to assess the clinical feasibility of using the telerehabilitation system in real life conditions (in the home environment), during an eight week period.

During their initial pulmonary rehabilitation session (held in the centre), participants will be offered to perform their pulmonary rehabilitation program at home, using the telerehabilitation system. Those who agree to participate will be taught to use the system during this first face-to-face session. The telerehabilitation system as well as a cycle ergometer will be subsequently provided in their home environment by a local home healthcare provider.

The telerehabilitation program will take place over an eight-week period and includes:

* Endurance exercise training on a cycle ergometer (performed independently with remote monitoring or through video conference (also with remote monitoring), according to the participant's preference), three times per weeks. The duration of the sessions along with the training intensity will be progressively adjusted using an automated algorithm (aimed to first increase the training duration up to forty-five minutes and then workload intensity). The algorithm is based on previous sessions performed, monitored data and perceived exertion.
* Peripheral muscle strengthening using the app (the patient will be requested to reproduce different exercises after watching a video) or through video conference, three times per weeks (thirty minutes).
* Daily walking (automated coaching based on Demeyer et al. Thorax. 2017).
* Self management education (one to nine sessions according to each individual's needs, scheduled through videoconference).
* A self evaluation of symptoms through daily or weekly questionnaires.

Different types of alerts will be triggered at the center according to remote monitoring : "non-adherence", "clinical issue" during endurance exercise sessions and change in "symptoms".

Participants will be encouraged to contact physiotherapists at the centre for any situation that would require assistance (related to their program or to cope with any technical issue).

ELIGIBILITY:
Inclusion Criteria:

* Age superior to eighteen years.
* Stable (> four weeks) chronic obstructive pulmonary disease, GOLD stage II to IV
* Referred to pulmonary rehabilitation (no contraindication to exercise training on a cycle ergometer).
* With or without oxygen during exercise.

Specific inclusion criteria for the first step of the study:

* Able to perform forty-five minutes of exercise training on a cycle ergometer.

Specific inclusion criteria for the second phase of the study:

* Person of legal age who may be present during home exercise sessions (relatives).

Non-inclusion Criteria:

* Pregnancy or likely to be.
* Guardianship.
* Unable to consent.
* Referred to pulmonary rehabilitation before lung cancer surgery.
* Referred to pulmonary rehabilitation before lung volume reduction surgery scheduled in the next few months.

Exclusion Criteria:

* Consent withdrawal

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Technical validity of the data transmitted remotely - pulse oximeter - concordance between datasets. | Data will be recorded immediately after the intervention.
  Comparison of paired datasets between the data recorded locally within the internal memory of the pulse oximeter and those collected from the telerehabilitation system.
Technical validity of the data transmitted remotely - physical activity tracker - concordance between datasets. | Data will be recorded immediately after the intervention.
  Comparison of paired dataset between the daily data, either automatically collected from the telerehabilitation system or self-reported by the participant (visually displayed on the physical activity tracker).
Technical validity of the data transmitted remotely - pulse oximeter - proportion of sessions transmitted. | Data will be recorded immediately after the intervention.
  The number of exercise sessions retrieved from the telerehabilitation system will be expressed in relation to the number of sessions performed.
Technical validity of the data transmitted remotely - physical activity tracker - proportion of sessions transmitted. | Data will be recorded immediately after the intervention.
  The number of days with physical activity data retrieved from the telerehabilitation system will be expressed in relation to the number of days that the tracker has been worn by the participant.
Technical validity of the data transmitted remotely - pulse oximeter - proportion of common usable data. | Data will be recorded immediately after the intervention.
  The proportion of data without artefacts will be compared between datasets. Artefacts will be identified for heart rate when values indicate two hundred fifty beats per minute and for transcutaneous oxygen saturation when values indicate hundred percent.
Technical validity of the data transmitted remotely - pulse oximeter - number of session required to be autonomous when using the system. | Data will be recorded immediately after the intervention.
  Participants will be taught to use the system and they will be requested to set data collection autonomously during the four next sessions. They will be considered autonomous when they will be able to set data collection autonomously without error. The number of sessions (after the first session) required to reach autonomy will be collected.

SECONDARY OUTCOMES:
Endurance exercise capacity - constant workload exercise testing. | Baseline and immediately after the intervention.
  Time to exhaustion (in second) during a constant workload exercise testing on a cycle ergometer at seventy-five percent of the maximal workload achieved during a previously performed incremental cardiopulmonary exercise testing.
Endurance exercise capacity - six-minute walking test. | Baseline and immediately after the intervention.
  Number of meters performed during the six-minutes walking test, performed in a thirty metre long corridor.
Endurance exercise capacity - six-minute stepper test. | Baseline and immediately after the intervention.
  Number of steps performed during the six-minutes stepper test.
Maximal voluntary isometric quadriceps force. | Baseline and immediately after the intervention.
  Data will be recorded using a handheld manometer.
Self-reported quality of life. | Baseline and immediately after the intervention.
  Saint George's Respiratory Questionnaire.
Functional dyspnea. | Baseline and immediately after the intervention.
  Modified Medical Research Council dyspnea scale.
Health status. | Baseline and immediately after the intervention.
  Chronic obstructive pulmonary disease Assessment Test.
Anxiety. | Baseline and immediately after the intervention.
  Hospital And Anxiety questionnaire - anxiety sub scale.
Depression. | Baseline and immediately after the intervention.
  Hospital And Anxiety questionnaire - depression sub scale.
Cognitive Function. | Baseline and immediately after the intervention.
  Montreal Cognitive Assessment test.
Objective physical activity. | Baseline and immediately after the intervention.
  Objective physical activity will be assessed using a physical activity tracker (different from the one used with the telerehabilitation system) and expressed as daily step count over a ten-day period. A given day will be considered as valid if the device is worn at least eight hours and the outcome will be considered as valid for a given participant if the measurement includes at least four valid week days.
Adherence - exercise training. | Data will be collected through study completion, an average of 8 weeks.
  Adherence will be assessed as the number of exercise training sessions performed in relation to the number of sessions prescribed.
Adherence - self-management education. | Data will be collected through study completion, an average of 8 weeks.
  Adherence will be assessed as the number of self-management education sessions performed in relation to the number of sessions prescribed.
Adherence - symptoms monitoring questionnaires. | Data will be collected through study completion, an average of 8 weeks.
  Adherence will be assessed as the number of days with fulfilled questionnaires relative to the number of days.
Use of the telerehabilitation system. | Data will be collected through study completion, an average of 8 weeks.
  Logs related to the different components of the programs will be retrieved from the telerehabilitation system (number of click to each component of the eight-week period).
Usability of the system. | Data will be collected immediately after the intervention.
  Usability of the system will be assessed using the System Usability Scale.
Satisfaction - standardized questionnaire. | Data will be collected immediately after the intervention.
  Satisfaction will be assessed using the Client Satisfaction Questionnaire-8.
Satisfaction - purpose designed survey. | Data will be collected immediately after the intervention.
  Satisfaction will be assessed using purpose designed surveys intended for participants, their relatives and healthcare professional in charge of telerehabilitation program (Lickert scale).
Emotional perception of the system. | Data will be collected immediately after the intervention.
  Emotional perception of the system will be assessed using Emocards.
Participant's flow. | Data will be collected immediately after the intervention.
  Participant's flow with the system will be assessed using the FKS scale from Rheinberg et al. (2003).
Motivation to participate in the program using the telerehabilitation system. | Data will be collected immediately after the intervention.
  Motivation will be assessed through a one hour semi-directed interview.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Bonnevie, PT, PhD, Principal Investigator — ADIR Association, Rouen University, Rouen, France; Antoine Cuvelier, MD, Prof, Study Chair — CHU-Hôpitaux de Rouen, Rouen, France.; Jean-François Muir, MD, Prof, Study Chair — ADIR Association, Rouen, France.; Francis-Edouard Gravier, PT, PhD, Study Chair — ADIR Association, Rouen, France.; Aurélie Vallée, PhD, Study Chair — CogSci, Rouen, France.; Michelle Leclerc, PT, MSc, Study Chair — Union des Kinésithérapeutes Respiratoires, Rouen, France.; Zoe McKeough, PT, Prof, Study Chair — Faculty of Medicine and Health, The University of Sydney, Sydney, New South Wales, Australia.
Locations (1):
- ADIR Association, Bois-Guillaume, ADIR Association, France